CLINICAL TRIAL: NCT03735056
Title: Providing Emotional Support Around the Point of Multiple Sclerosis Diagnosis (PrEliMS): A Feasibility Randomised Controlled Trial
Brief Title: The PrEliMS Feasibility Trial
Acronym: PrEliMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Multiple Sclerosis Society UK (Unknown); Swansea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18053
Record Dates: First submitted 2018-09-21; First posted 2018-11-08 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: Diagnosis; Emotional support; Peer support
MeSH Terms: conditions — Multiple Sclerosis; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Usual care) (No Intervention): Receives usual care only.
- Group 2 (Usual care plus Support 1) (Experimental): Receives usual care plus Support 1 (MS Nurse Support) which includes one one-to-one, face-to-face session with an MS Nurse Specialist in a hospital setting (or via Skype). The session will include answering newly diagnosed patients' questions about MS, providing psychoeducation and teaching Acceptance and Commitment strategies (Hayes, Strosahl & Wilson, 1999), and referring to other services (based on needs). Participants will also be given a self-help workbook ('Better living with a diagnosis of MS: Patient Workbook') by the nurses. This session will take place within 2 weeks of diagnosis and last up to 90 minutes. It will be supplemented by phone calls (depending on participant needs). MS Nurses will receive training and on-going supervision from experienced clinical psychologists.
  Interventions: Other: MS Nurse Support
- Group 3 (Usual care plus Support 2) (Experimental): Receives usual care plus Support 2 (i.e. MS Nurse Support plus Peer Support). In addition to receiving the MS Nurse Support (i.e. Support 1, as described in Group 2), this group will also receive peer support which will be provided by Peer Support Workers who are patients/carers with lived experience and who are recruited and trained to deliver peer support under supervision from experienced clinical psychologists. It will be delivered one-to-one, face-to-face (in a community setting or via Skype, based on participants' preferences). Patients in this group will be triaged to a Peer Support Worker by the MS Nurse during the 2-week MS Nurse Support session. The sessions will be scheduled to a convenient time between weeks 2-6 after diagnosis and each session will last up to 60 minutes.
  Interventions: Other: MS Nurse Support; Other: Peer Support

INTERVENTIONS:
Other: MS Nurse Support — MS Nurse Support intervention is multi-faceted, involving various components (i.e. information provision and emotional support), and a range of strategies and techniques (e.g. psychoeducation, acceptance and commitment), delivered by MS Nurse Specialists, to provide standardised support and advice to patients at diagnosis, to establish and sustain coping strategies. MS Nurse Support intervention is person-centred and tailored to the needs and lifestyle of each participant.
  Arms: Group 2 (Usual care plus Support 1); Group 3 (Usual care plus Support 2)
Other: Peer Support — Peer Support will be delivered by Peer Support Workers using information provision and supportive listening to provide support and advice to patients at diagnosis, and to provide patients the opportunity to talk freely, extensively and confidentially about their experiences, thoughts and feelings about MS diagnosis and its effects on their lives in a non-judgmental and safe environment. Peer Support intervention is person-centred and tailored to the needs and lifestyle of each participant.
  Arms: Group 3 (Usual care plus Support 2)

SUMMARY:
The PrEliMS study is a mixed-methods feasibility randomised controlled trial of a point of diagnosis intervention programme which aims to provide emotional support for newly diagnosed people with Multiple Sclerosis (MS). This feasibility study will enable us to plan for a definitive trial to evaluate the clinical and cost-effectiveness of this point of diagnosis intervention programme. The aim is to assess the feasibility of the trial procedures and intervention, and to evaluate the key feasibility parameters before proceeding to a definitive trial. Participants (N=60) will be randomised into three groups: (1) usual care; (2) usual care + Support 1 (MS Nurse Support); (2) usual care + Support 2 (MS Nurse Support plus Peer Support).

DETAILED DESCRIPTION:
Potential participants will be people who have been recently diagnosed with MS (or currently going through diagnosis process), and who are aged 18 years or over, recruited through MS clinics. Participants, after consent, will complete baseline measures before being randomised into to one of three groups: (1) usual care; (2) usual care + Support 1 (MS Nurse Support); (2) usual care + Support 2 (MS Nurse Support plus Peer Support). Group 1 (20 patients) will not receive any intervention. Group 2 (20 patients) will receive Support 1 which will include one face-to-face support session delivered by an MS Nurse. Group 3 (20 patients) will receive Support 2 which includes MS Nurse Support (i.e., Support 1) plus Peer Support. Peer Support will include a minimum of two peer support session delivered by Peer Support Workers (i.e. patients with lived experiences). All groups will receive usual care. The outcome measures will be collected at 3 and 6 months after randomisation by all participants. Feedback interviews with up to 21 participants (7 from each group) and up to 10 service providers (5 MS Nurses who delivered the MS Nurse Support and 5 Peer Support Workers who delivered the Peer Support) will be conducted to assess what parts of the intervention were helpful or unhelpful, the acceptability of randomisation and trial procedures, and the appropriateness of the measures used.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible to join the trial if they:

* are 18 years or over
* have recently received a diagnosis of MS (any type of MS) or currently going through MS diagnosis process)
* can communicate in English
* able and willing to give consent
* not receiving psychological intervention

Exclusion Criteria:

Patients will be excluded if they:

* have a severe co-morbid psychiatric condition (e.g. dementia), as reported by patients or their carers or confirmed by the clinical team making the initial approach
* are currently receiving psychological interventions or received this within the last three months (we will not exclude those on medication for their mood problems but will record this information).
* do not have mental capacity to consent to take part in the trial
* are unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of trial procedures | Daily throughout data collection
  [Note: As feasibility studies are used to estimate important parameters to inform the design of a full trial (NIHR, 2018), we outline the key outcomes related to feasibility. These are described below. Please see Outcome 1-15.]
  Feasibility of trial procedures will be assessed through feedback interview (qualitative) data from participants and service providers (i.e., questions about the research process/procedures, and suggested changes to the study).
Acceptability of trial procedures | Daily throughout data collection
  Assessed through feedback interview (qualitative) data from participants and service providers on the trial procedures.
Feasibility of randomisation protocol | Daily throughout data collection
  Assessed through feedback interview (qualitative) data on randomisation protocol and willingness and acceptance of patients to be randomised.
Feasibility of recruitment | Daily throughout data collection
  Number of those eligible who expressed interest/discussed with researcher, number of consenting/randomised patients, reasons for non-participation, retention rates, feedback interview (qualitative) data.
Estimating sample size needed for a Phase III RCT | Daily throughout data collection
  Sample size calculated through effect sizes from ANOVAs, standard deviations and attrition rates.
Appropriateness of measures | Daily throughout data collection
  Completion rates of outcome measures, number of missing online and postal data, estimates of time (minutes) taken to complete measures (from online/phone data or feedback interview data).
Feasibility of self-report data collection | Daily throughout data collection
  Number of missing online and postal data
Feasibility of audio recording support sessions | Daily throughout data collection
  Number of participants consenting to audio recording of sessions and feedback interview data
Acceptability of interventions (Support 1 and Support 2) | Daily throughout intervention delivery
  Drop-out rates (and reasons for withdrawal), number of Support 1 and Support 2 sessions completed, feedback interview data.
Feasibility of delivering Support 1 intervention | Daily throughout intervention delivery
  Number of missed and rescheduled sessions, length of sessions (minutes), operational issues in delivering intervention through feedback interview data.
Feasibility of delivering Support 2 intervention | Daily throughout intervention delivery
  Number of missed and rescheduled sessions, length of sessions (minutes), operational issues in delivering intervention through feedback interview data.
Credibility of interventions | Daily throughout data collection
  Assessed through qualitative feedback interview data (i.e., questions about the content of the intervention, changes experienced).
Fidelity of intervention | Daily throughout intervention delivery
  Fidelity rating on audio data from a sample of support sessions against criteria for PrEliMS model consistency.
Documentation of usual care | Daily throughout data collection
  Data obtained through service use questionnaire and feedback interviews.
Feasibility of collecting data for an economic evaluation using a bespoke service use questionnaire | Daily throughout data collection
  Number of missing or clearly invalid service use questionnaire data, completion rates, exploration of possible ceiling effects, feedback interview (qualitative) data.

OTHER OUTCOMES:
Perceived stress | Baseline, 3-month follow-up, and 6-month follow-up
  Perceived Stress Scale 4 (PSS4; Cohen, Kamarck, & Mersmelstein, 1983; Cohen & Williamson, 1988) to measure the level of perceived stress among people with MS by assessing their level of perceived uncontrollability and unpredictability on a 5 point scale (0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often). The scores for each question are added (after reverse scoring two of the four questions) to give a total score ranging from 0 to 16, with higher scores indicating higher stress.
Mood | Baseline, 3-month follow-up, and 6-month follow-up
  Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983) will be used to measure the level of mood disturbances. It is a 14-item scale and each item is scored from 0 to 3. The total scores range from 0 to 21 for the anxiety subscale and also for the depression subscale, with higher scores indicating greater levels of anxiety or depression.
Psychological impact of MS | Baseline, 3-month follow-up, and 6-month follow-up
  Multiple Sclerosis Impact Scale 29 (MSIS-29) - psychological subscale (Rasch, version 2; Hobart, Lamping, Fitzpatrick, Riazi, & Thompson, 2001; Ramp, Khan, Misajon, & Pallant, 2009) will be used to assess the perceived psychological impact of MS. Psychological subscale has 9 items with 4-point response categories for each item ("not at all", "a little", "moderately", "extremely"). The total score range from 9 to 36, with lower scores indicating little impact of MS and higher scores indicating greater impact.
Self-efficacy | Baseline, 3-month follow-up, and 6-month follow-up
  Multiple Sclerosis Self-efficacy Scale (MSSE; Rigby, Domenech, Thornton, Tedman, & Young, 2003) will be used to assess the extent to which participants feel in control of their condition. The scale has 14 items. Each item is presented with a 6-point Likert scale, ranging from "Strongly Disagree" to "Strongly Agree". The scores for each item are added (after reverse scoring six of the 14 items) to give a total score ranging from 14-84, with higher scores indicating an elevated level of self-efficacy.
Health-related quality of life | Baseline, 3-month follow-up, and 6-month follow-up
  EQ-5D-5L (Herdman et al., 2011) will be used as a generic patient-reported measure of health-related quality of life and to derive health utilities.
Service use questionnaire | Baseline, 3-month follow-up, and 6-month follow-up
  Service use questionnaire was adapted from the service use questionnaire used in the CRAMMS trial (Lincoln et al. 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Roshan das Nair, PhD, Principal Investigator — University of Nottingham; Gogem Topcu, PhD, Study Director — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No